CLINICAL TRIAL: NCT04117256
Title: Effectiveness of Transcranial and Suboccipital Direct Current Stimulation on Endogenous Pain Modulation System in Healthy Volunteers.
Brief Title: Transcranial Versus Suboccipital Direct Current Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Universidad Rey Juan Carlos (Other); Hospital Nacional de Parapléjicos de Toledo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GuillermoGB; 0220493 (Registry Identifier: Guillermo García Barajas)
Record Dates: First submitted 2019-09-30; First posted 2019-10-07 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Pain; Transcranial Direct Current Stimulation
Keywords: Direct Current Stimulation; Conditioned Pain Modulation; Endogenous Pain Modulation; Temporal Summation; Pressure Pain Threshold; Pain
MeSH Terms: conditions — Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Paralled randomized controlled trial with cross-control design. Two groups of subjects will be randomly selected, a Transcranial stimulation group and a suboccipital stimulation group. Each group will perform two intervention sessions in a randomized order, a session with direct current stimulation and a sham stimulation session.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding of the assessor: all the assessments will be made by a different researcher who apply all the interventions. Assessor will not have vision of the place where the electrodes are located neither the parameters used.
  Blinding of the subjects: Although subjects will be blinded to the hypothesis of the study, the transcranial and suboccipital location of the electrodes cannot be blinded. Direct current and sham stimulation will be blinded. For the sham condition subjects will feel the stimulation sensation for 30 seconds and then the stimulator will turn off. The same equipment, identical electrodes, and cables will be used. In addition, subjects will not have a view of the computer screen.
  Blinding of the person who apply the intervention: Although transcranial and suboccipital conditions cannot be blinded. The direct current and sham stimulation will be apply by the blind-mode of the stimulator using locking codes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcranial Stimulation (Active Comparator): Transcranial stimulation on the primary motor cortex (M1) with anode located on the point C3 (10/20 EEG system), and the cathode on contralateral supraorbital zone.
  Interventions: Device: Direct Current Stimulation; Device: Sham DCS
- Suboccipital Stimulation (Active Comparator): Suboccipital stimulation with anode located at the upper cervical level and cathode was placed on the lateral part of right shoulder.
  Interventions: Device: Direct Current Stimulation; Device: Sham DCS

INTERVENTIONS:
Device: Direct Current Stimulation — 20 minutes of direct current stimulation using an intensity of 1.5mA and electrode size of 6x4cm
Device: Sham DCS — 20 minutes of sham stimulation. Subjects will be stimulated during the first 30 seconds. After that, a ramp down of 10 seconds and then the stimulator is turned-off.

SUMMARY:
Randomized controlled trial, in parallel with cross-control design. Two groups of healthy subjects will be randomly selected to transcranial stimulation group or suboccipital stimulation group. Each group receive in a randomized order a real direct current session and a sham session. The study is based on the hypothesis that the application of direct current sitmulation applied at the suboccipital level produce higher modifications on endogenous pain modulation system than transcranial stimulation.

DETAILED DESCRIPTION:
The development of the project will be based on the Declarations of the World Medical Association of Helsinki. Every subject will be informed about the nature of the study, willingness to participate, the proposed objectives, as well as possible adverse effects that may occur in its implementation. Every subject will be asked to give their signed consent to participate in the study. The study will be suspended at any time, if the patient wishes.

Healthy volunteers will be recruited from the city of Toledo, between the ages of 18 and 40. The detection and selection of the sample will be carried out between the students of the University of Castilla-La Mancha and personnel of the Hospital Nacional de Parapléjicos who meet the inclusion criteria and give their consent voluntarily to participate in the study.

The calculation of the sample size will be carried out using the G * Power software program (version 3.1), for clinical studies with two intervention groups. Conditioned pain modulation will be chosen as the primary outcome variable. Assuming an α level of 0.05 and a statistical power of 85%, with a moderate effect size for the ANOVA test (0.25).

The experiment will be carried out in the clinical laboratory of the Sensory-Motor Function Research Group of the Hospital Nacional de Parapléjicos. Under attenuated sound conditions, and at a stable temperature in the range of (22 °C-26 °C).

In the first session of the study, a small interview will be carried out to determine if there is any exclusion criterion. The initial measurements will consist of sociodemographic variables and psychological variables, which will then be used to categorize groups and analyze covariates. A parallel randomized controlled trial with cross-control design is proposed. Two groups of healthy subjects will be randomly selected to transcranial direct current stimulation (DCS) group or suboccipital DCS group. Each group receive in a randomized order and with a double blind design a real direct current session and a sham session. An assessment is made before and after each intervention.

Subjects will remain in a sitting position, with their backs resting in a relaxed position. In all interventions a direct current stimulator (DC-stimulator, Neuroconn) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years.
* Healthy volunteers (without neurological injury and no history of pain in the last 6 months).
* Ability to perform all clinical test and understand the process of the study, as well as obtaining informed consent.
* Tolerance to the application of electrotherapy.

Exclusion Criteria:

* Previous history of surgical intervention at the cervical level.
* Have been treated with an electric current similar to that applied prior to the intervention.
* Sensitivity altered in the area of application of the intervention.
* No commitment to continuity.
* History of neuromuscular disease.
* Epilepsy.
* Injuries, surgery or pain affecting the upper limb.
* Material of osteosynthesis at the cervical level.
* Diabetes.
* History of cancer.
* Cardiovascular disease.
* Presence of pacemakers or any other implanted electrical device.
* Take medication during the study and in the 7 days prior to the study.
* Consumption of narcotic substances during the study and in the 7 days prior to the study.
* Presence of tattoos or any other external agent introduced in the treatment and assessment area (hand).
* Pregnancy.
* Presence of severe and frequent headaches.
* Ulcers or scars in the skin at the location of the electrodes

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Conditioned Pain Modulation | Baseline at 0 min
  For this protocol the test stimulus (TS) and the conditioning stimulus (CS) will be applied sequentially (first CS, followed by TS), heterotopic, and contralateral. The CS temperature will be 12 °C on the cold pressor test to induce a perception of pain. The subjects will have to submerge the non-dominant hand in the cold water bath for 30s, and evaluate the CS-induced pain intensity at 10, 20, and 30s (t1, t2 and t3 respectively). After assessing CS-induced pain intensity at the 30s of immersion participants will withdraw their hand from the water bath, and will have to fix their attention to the dominant hand where TS was immediately applied. The TS-induced pain assessment at 10, 20, and 30s (t1, t2 and t3).
Change from baseline Conditioned Pain Modulation | At 30 min
  For this protocol the test stimulus (TS) and the conditioning stimulus (CS) will be applied sequentially (first CS, followed by TS), heterotopic, and contralateral. The CS temperature will be 12 °C on the cold pressor test to induce a perception of pain. The subjects will have to submerge the non-dominant hand in the cold water bath for 30s, and evaluate the CS-induced pain intensity at 10, 20, and 30s (t1, t2 and t3 respectively). After assessing CS-induced pain intensity at the 30s of immersion participants will withdraw their hand from the water bath, and will have to fix their attention to the dominant hand where TS was immediately applied. The TS-induced pain assessment at 10, 20, and 30s (t1, t2 and t3).

SECONDARY OUTCOMES:
Baseline Temporal Summation | At 5 min
  For the evaluation of the habituation and temporal summation of pain, heat stimuli of a "p-3" intensity without conditioning stimulus (CS) will be applied. The tonic heat stimulus will be applied on the surface of the tenar eminence of the dominant hand by 8 consecutive stimuli separated from each other by 1.5 seconds, evaluating the pain perceived during the first and the eighth stimulus, and at 15 seconds after the stimulation. The temperature will be determined individually, in order to reflect the general level of discomfort that the stimulus could produce according to the visual analog scale (0-10).
Change from baseline Temporal Summation | At 35 min
  For the evaluation of the habituation and temporal summation of pain, heat stimuli of a "p-3" intensity without conditioning stimulus (CS) will be applied. The tonic heat stimulus will be applied on the surface of the tenar eminence of the dominant hand by 8 consecutive stimuli separated from each other by 1.5 seconds, evaluating the pain perceived during the first and the eighth stimulus, and at 15 seconds after the stimulation. The temperature will be determined individually, in order to reflect the general level of discomfort that the stimulus could produce according to the visual analog scale (0-10).
Baseline Pressure Pain Threshold | at 10 min
  To record the mechanical pain threshold, a point will be marked on the Tibialis Anterior muscle and on the dorsal surface of the right hand, specifically on the second metacarpal lateral border, approximately 3 cm proximal to the interdigital fold. This zone is especially sensitive to pressure. For registration, the digital algometer with 0.1 N increment scale (Wagner Instruments brand, model FDIX), with a circular applicator of 1 cm in diameter will be used. Once the applicator is placed perpendicular to the skin, the pressure will increase at a rate of approximately 5 N / s. Three measures will be taken with an interval between measures of 10 seconds, the average of the three measurements will be taken as threshold of pain to the pressure.
Change from baseline Pressure Pain Threshold | at 40 min
  To record the mechanical pain threshold, a point will be marked on the Tibialis Anterior muscle and on the dorsal surface of the right hand, specifically on the second metacarpal lateral border, approximately 3 cm proximal to the interdigital fold. This zone is especially sensitive to pressure. For registration, the digital algometer with 0.1 N increment scale (Wagner Instruments brand, model FDIX), with a circular applicator of 1 cm in diameter will be used. Once the applicator is placed perpendicular to the skin, the pressure will increase at a rate of approximately 5 N / s. Three measures will be taken with an interval between measures of 10 seconds, the average of the three measurements will be taken as threshold of pain to the pressure.

OTHER OUTCOMES:
State-Trait Anxiety Questionnaire (STAI-ES) | At 0 min
  We will use the adapted version to the Spanish of the State Scale (STAI-ES) of the "State-Trait Anxiety Questionnaire" (STAI). The STAI is a well-known scale of self-report, comprising two self-assessment subscales that measure two concepts of anxiety: state (S) and trait (T). It is composed of 40 items with 4 possible answers each (score 0 to 3). The total scores for each of the subscales range from 0 to 60 points. Specifically STAI-ES evaluates the anxiety-state in a great variety of situations.
Beck Depression Inventory (BDI). | At 0 min
  Most commonly used questionnaire at the global and national levels to assess depression. We will use the adaptation to the Spanish of the Beck II depression inventory. It consists of 21 items to measure the affective, cognitive situation and the signs and symptoms of depression during the last two weeks. High scores indicate high levels of depressive symptoms. This inventory has demonstrated excellent psychometric properties

CONTACTS AND LOCATIONS:
Overall Officials: Julian Scott Taylor, Physiology, Study Director — Hospital Nacional de Parapléjicos de Toledo
Locations (1):
- Hospital Nacional de Parapléjicos de Toledo, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No
Data will be shown if requested

REFERENCES:
- [Background] Klein MM, Treister R, Raij T, Pascual-Leone A, Park L, Nurmikko T, Lenz F, Lefaucheur JP, Lang M, Hallett M, Fox M, Cudkowicz M, Costello A, Carr DB, Ayache SS, Oaklander AL. Transcranial magnetic stimulation of the brain: guidelines for pain treatment research. Pain. 2015 Sep;156(9):1601-1614. doi: 10.1097/j.pain.0000000000000210. PMID 25919472
- [Background] O'Connell NE, Wand BM, Marston L, Spencer S, Desouza LH. Non-invasive brain stimulation techniques for chronic pain. Cochrane Database Syst Rev. 2010 Sep 8;(9):CD008208. doi: 10.1002/14651858.CD008208.pub2. PMID 20824873
- [Background] Brunoni AR, Amadera J, Berbel B, Volz MS, Rizzerio BG, Fregni F. A systematic review on reporting and assessment of adverse effects associated with transcranial direct current stimulation. Int J Neuropsychopharmacol. 2011 Sep;14(8):1133-45. doi: 10.1017/S1461145710001690. Epub 2011 Feb 15. PMID 21320389
- [Background] Brunoni AR, Nitsche MA, Bolognini N, Bikson M, Wagner T, Merabet L, Edwards DJ, Valero-Cabre A, Rotenberg A, Pascual-Leone A, Ferrucci R, Priori A, Boggio PS, Fregni F. Clinical research with transcranial direct current stimulation (tDCS): challenges and future directions. Brain Stimul. 2012 Jul;5(3):175-195. doi: 10.1016/j.brs.2011.03.002. Epub 2011 Apr 1. PMID 22037126
- [Background] Albu S, Gomez-Soriano J, Avila-Martin G, Taylor J. Deficient conditioned pain modulation after spinal cord injury correlates with clinical spontaneous pain measures. Pain. 2015 Feb;156(2):260-272. doi: 10.1097/01.j.pain.0000460306.48701.f9. PMID 25599447
- [Background] Yarnitsky D. Role of endogenous pain modulation in chronic pain mechanisms and treatment. Pain. 2015 Apr;156 Suppl 1:S24-S31. doi: 10.1097/01.j.pain.0000460343.46847.58. PMID 25789433
- [Background] Staud R, Weyl EE, Riley JL 3rd, Fillingim RB. Slow temporal summation of pain for assessment of central pain sensitivity and clinical pain of fibromyalgia patients. PLoS One. 2014 Feb 18;9(2):e89086. doi: 10.1371/journal.pone.0089086. eCollection 2014. PMID 24558475
- [Background] Pud D, Granovsky Y, Yarnitsky D. The methodology of experimentally induced diffuse noxious inhibitory control (DNIC)-like effect in humans. Pain. 2009 Jul;144(1-2):16-9. doi: 10.1016/j.pain.2009.02.015. Epub 2009 Apr 8. No abstract available. PMID 19359095
- [Background] Nussbaum EL, Downes L. Reliability of clinical pressure-pain algometric measurements obtained on consecutive days. Phys Ther. 1998 Feb;78(2):160-9. doi: 10.1093/ptj/78.2.160. PMID 9474108
- [Background] Sanz J, García-Vera MP, Espinosa R, Fortún M, Vázquez C. Adaptación española del Inventario para la Depresión de Beck-II (BDI-II): 3. Propiedades psicométricas en pacientes con trastornos psicológicos. Clínica y Salud. 2005;16(2):121-42.
- [Background] Spielberger CD. Manual for the State-Trait Anxiety Inventory (STAI Form Y). Consult Psychol Palo Alto. 1983;4-6.
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Fregni F, Boggio PS, Lima MC, Ferreira MJ, Wagner T, Rigonatti SP, Castro AW, Souza DR, Riberto M, Freedman SD, Nitsche MA, Pascual-Leone A. A sham-controlled, phase II trial of transcranial direct current stimulation for the treatment of central pain in traumatic spinal cord injury. Pain. 2006 May;122(1-2):197-209. doi: 10.1016/j.pain.2006.02.023. Epub 2006 Mar 27. PMID 16564618